CLINICAL TRIAL: NCT06003231
Title: A Phase 2 Basket Study of Disitamab Vedotin in Adult Subjects With Previously Treated, Locally-Advanced Unresectable or Metastatic Solid Tumors That Express HER2
Brief Title: A Study of Disitamab Vedotin in Previously Treated Solid Tumors That Express HER2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNDV-005; C5731005 (Other: Alias Study Number); 2023-504445-31-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms
Keywords: NSCLC; Ovarian Cancer; Endometrial Cancer; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms | interventions — disitamab vedotin; RC48 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Head and neck cancer (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Non-small cell lung cancer (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Ovarian cancer (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Endometrial cancer (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin

INTERVENTIONS:
Drug: disitamab vedotin — Given into the vein (IV, intravenous) every 2 weeks
  Other Names: RC48, RC48-ADC

SUMMARY:
This clinical trial is studying advanced or metastatic solid tumors. Once a solid tumor has grown very large in one spot or has spread to other places in the body, it is called advanced or metastatic cancer. Participants in this study must have head and neck cancer, non-small cell lung cancer, endometrial cancer, or ovarian cancer. In the first part of the study, participants must have tumors that have a marker called HER2.

This clinical trial uses an experimental drug called disitamab vedotin (DV). DV is a type of antibody-drug conjugate or ADC. ADCs are designed to stick to cancer cells and kill them. In this study, all participants will get DV once every 2 weeks.

This study is being done to see if DV works to treat different types of solid tumors that express HER2. It will also test how safe the drug is for participants. This trial will also study what side effects happen when participants get the drug. A side effect is anything a drug does to your body besides treating the disease.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Head and neck cancer (HNC)

  * Must have pathologically-documented carcinoma of the head and neck with primary tumor site arising from the oral cavity, salivary gland, oropharynx, hypopharynx, and larynx; tumors arising from the nasopharynx are excluded.
  * Unresectable locally recurrent or metastatic stage disease
  * Prior therapies:

    * Participants must have disease progression after treatment with a platinum-based therapy
* Cohort 2: Non-small cell lung cancer (NSCLC)

  * Pathologically documented NSCLC
  * Unresectable locally-advanced or metastatic stage disease
  * Prior therapies

    * Must have progressed during or after a platinum-based therapy for LA/metastatic disease or, within 6 months of platinum-based adjuvant, neoadjuvant, or concomitant chemoradiotherapy for early or locally-advanced stage disease
    * Must have received prior anti-PD(L)1 therapy, unless contraindicated
    * Participants with known AGAs must have received appropriate targeted therapy, where available.
    * No more than 2 prior lines of cytotoxic chemotherapy for advanced disease
* Cohort 3: Ovarian Cancer

  * Pathologically documented epithelial cancers of ovarian, fallopian tube, or peritoneal origin
  * Unresectable locally-advanced or metastatic stage disease
  * Prior therapies

    * Must have platinum resistant disease (6 months or less between the completion of platinum-based treatment and identification of recurrence)
    * Must not have received more than 4 lines of prior cytotoxic chemotherapies for advanced disease
    * Participants with known BRCA mutations are permitted, but participants must have received targeted therapy with a PARP inhibitor
    * May have received prior anti-PD(L)1 therapy
* Cohort 4: Endometrial Cancer

  * Must have pathologically documented adenocarcinoma of the endometrium
  * Must have unresectable locally-advanced or metastatic stage disease.
  * Prior therapies

    * Must have relapsed/progressed after at least one prior platinum-based chemotherapy for recurrent, metastatic or primary unresectable disease
    * Must not have received more than 3 lines of prior cytotoxic chemotherapies for advanced disease
    * May have received prior anti-PD(L)1 therapy
* HER2 expression of 1+, 2+, or 3+, as determined by local IHC testing on a fresh or archival tumor tissue. Note: Participants with HER2 mutations are eligible.
* Measurable disease per RECIST v1.1 criteria as assessed by the investigator
* Able to provide formalin-fixed, paraffin-embedded (FFPE) tumor tissue blocks (or freshly sectioned slides)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Prior treatment with an MMAE-containing agent.
* Known hypersensitivity to any excipient contained in the drug formulation of disitamab vedotin.
* History of another invasive malignancy within 2 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
* Active untreated CNS or leptomeningeal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) per Response Evaluation in Solid Tumors version 1.1 (RECIST v1.1) by investigator assessment | Approximately 3 years
  The proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the investigator

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after the last dose of DV; approximately 5 years
  Any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratories abnormalities | Through 30-37 days after the last dose of DV; approximately 5 years
Number of participants with dose alterations due to AEs | Approximately 5 years
Confirmed Disease Control Rate (DCR) per RECIST v1.1 by investigator assessment | Approximately 5 years
  The proportion of participants with stable disease (SD) or confirmed CR or PR according to RECIST v1.1
Duration of Response (DOR) per RECIST v1.1 by investigator assessment | Approximately 5 years
  The time from start of the first documentation of objective tumor response of CR or PR (that is subsequently confirmed) to the first documentation of progressive disease (PD) per RECIST v1.1, or to death due to any cause
Progression free survival (PFS) per RECIST v1.1 by investigator assessment | Approximately 5 years
  PFS is defined as the time from the start of study treatment to the first documentation of PD per RECIST v1.1 or death due to any cause, whichever occurs first
Overall Survival (OS) | Approximately 5 years
  The time from the start of study treatment to the date of death due to any cause
Pharmacokinetic (PK) parameter - Area under the concentration-time curve to the time of the last quantifiable concentration (AUClast) | Approximately 1 month
  Analyzed through cycle 2.
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after the last dose of DV; approximately 5 years
  Analyzed through end of treatment.
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after the last dose of DV; approximately 5 years
  Analyzed through end of treatment.
Incidence of antidrug antibodies (ADAs) | Through 30-37 days after the last dose of DV; approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- United States (72):
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Chandler, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Gilbert, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Glendale, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Mesa, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Phoenix, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Scottsdale, Arizona
  - Valkyrie Clinical Trials(Additional Suite), Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Davis Comprehenvise Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Providence Medical Foundation, Santa Rosa, California
  - PCM Trials, Denver, Colorado
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital-Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Trumbull, Trumbull, Connecticut
  - Sylvester Comprehensive Cancer Center- The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Hospital and Clinics Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Kendall, Miami, Florida
  - Sylvester Comprehensive Cancer Center Plantation, Plantation, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Wellstar MCG Health Clinical Research Pharmacy, Augusta, Georgia
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Minnesota Oncology Hematology, P.A., Burnsville, Minnesota
  - Allina Health Cancer institute, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A., Coon Rapids, Minnesota
  - M Health Fairview Cancer Clinic-Edina, Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Fridley, Minnesota
  - Minnesota Oncology Hematology, P.A., Maple Grove, Minnesota
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A., Maplewood, Minnesota
  - Allina Health Cancer Institute (Virginia Piper Cancer Institute), Minneapolis, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Health Cancer Center, Robbinsdale, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regulatory location : MMCORC, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Allina Health Cancer Institute-United(VPCI), Saint Paul, Minnesota
  - Minnesota Oncology Hematology, P.A. Cornerstone Medical Specialty Center, Woodbury, Minnesota
  - Optimum Clinical Research Group, LLC, Albuquerque, New Mexico
  - Southwest Women's Oncology Inc, Albuquerque, New Mexico
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Hospital-Long Island, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center At NYU Langone, New York, New York
  - Laura & Issac Perlmutter Cancer Center-NYU Ambulatory Care Center(ACC), New York, New York
  - NYU Langone Hospitals, NYU Langone Rusk Ambulatory Surgical Pharmacy, New York, New York
  - NYU Langone Hospitals, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - Duke University Medical Center, Investigational Chemotherapy Services, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - Providence St. Vincent Medical Center- Investigational Drug Services, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish First Hill IDS Pharmacy, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University Clinical Trials Unit., Macquarie University, New South Wales
  - Macquarie University Clinic, Macquarie University, New South Wales
  - Macquarie University Hospital Pharmacy, Macquarie University, New South Wales
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Baxter Healthcare, Old Toongabie, New South Wales
  - Peninsula & South Eastern Hematology and Oncology Group (PASO), Frankston, Victoria
  - Blacktown Hospital, Blacktown
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Centre Intégré de Cancérologie du CHU de Québec-Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
- Fondazione IRCCS San Gerardo dei Tintori., Monza (MB), Monza and Brianza, Italy
- South Korea (3):
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario Reina Sofia, Córdoba
  - Hospital Provincial, Córdoba
  - Clinica Universidad de Navarra Madrid, Madrid
- United Kingdom (3):
  - The Royal Marsden NHS Foundation Trust (RM), Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust (RM), London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNDV-005